CLINICAL TRIAL: NCT00618540
Title: Reduced Intensity Hematopoietic Cell Transplantation for Patients With Resistant Langerhans Cell Histiocytosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007UC002; UMN-0612M98407 (Other: IRB, University of Minnesota); LCH-HCT-2006 (Other: Histiocyte Society); UMN-MT2006-07 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2008-02-19; First posted 2008-02-20 (Estimated); Results first posted 2015-11-03 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Histiocytosis, Langerhans-cell
Keywords: childhood Langerhans cell histiocytosis
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — Alemtuzumab; fludarabine phosphate; Melphalan; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab (Experimental): Patients administered with alemtuzumab, fludarabine phosphate, melphalan and donor stem cell transplantation in children with resistant Langerhans cell histiocytosis.
  Interventions: Biological: alemtuzumab; Drug: fludarabine phosphate; Drug: melphalan; Procedure: stem cell transplantation

INTERVENTIONS:
Biological: alemtuzumab — Administered intravenously (IV) 0.2 mg/kg on Days -8 through -4.
  Other Names: Campath(R)
Drug: fludarabine phosphate — Administered 30 mg/m2 intravenously (IV) over 30-60 min on Days -7 through -3. (dose adjust if age <12 months)
  Other Names: Fludara(R)
Drug: melphalan — Administered 140 mg/m2 intravenously (IV) over 30 min on Day -2 (dose adjust if age <12 months)
  Other Names: Alkeran
Procedure: stem cell transplantation — Administered as allogeneic hematopoietic, peripheral blood or umbilical cord blood transplantation
  Other Names: Stem cell transplant

SUMMARY:
RATIONALE: Giving a monoclonal antibody, such as alemtuzumab, and chemotherapy drugs, such as fludarabine and melphalan, before a donor stem cell transplant helps stop the patient's immune system from rejecting the donor's stem cells and helps stop the growth of abnormal cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil before and after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving alemtuzumab together with fludarabine and melphalan followed by a donor stem cell transplant works in treating young patients with resistant Langerhans cell histiocytosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the overall and disease-free survival of poor-risk pediatric patients with Langerhans cell histiocytosis at 1 and 3 years after reduced-intensity hematopoietic cell transplantation (RI-HCT).

Secondary

* To determine day 100 transplantation-related mortality.
* To determine the incidence of hematopoietic recovery and chimerism at day 100 and at 1 year post RI-HCT.
* To determine the incidence of grades II-IV and III-IV acute graft-versus-host disease (GVHD).
* To determine the incidence of chronic GVHD.

OUTLINE: This is a multicenter study.

* Non-myeloablative conditioning: Patients receive alemtuzumab intravenously (IV) over 2 hours on days -8 to -4, fludarabine phosphate IV over 30-60 minutes on days -7 to -3, and melphalan IV over 15-30 minutes on day -2. Some patients may receive anti-thymocyte globulin IV on days -6 to -2 instead of alemtuzumab.
* Graft-versus-host disease prophylaxis and immunosuppression: Patients receive cyclosporine A (CSA) IV or orally 2-3 times daily beginning on day -3 and continuing until day 50 post transplantation, followed by a taper over 8 weeks in the absence of GVHD or donor lymphocyte infusion given for decreasing donor chimerism. Patients with mismatched donors (any source) and those receiving peripheral blood stem cells also receive mycophenolate mofetil (MMF) IV or orally 2-3 times daily beginning on day -3 and continuing to day 30 or 7 days after engraftment, whichever day is later, in the absence of GVHD. In patients with acute GVHD requiring systemic therapy, Mycophenolate mofetil (MMF) may be stopped 7 days after initiation of systemic therapy.
* Allogeneic hematopoietic stem cell infusion: Patients undergo infusion of bone marrow (preferred) or peripheral blood stem cells on day 0. Patients also receive filgrastim (G-CSF) subcutaneously or IV beginning on day 8 and continuing until blood counts recover for 2 consecutive days.
* Donor lymphocyte infusion (DLI): Patients with mixed chimerism (i.e., < 95% donor) and those with < 50% donor T-cell engraftment at any engraftment assessment time point are eligible for DLI, in the absence of GVHD. If mixed chimerism persists, escalating doses of CD3-positive lymphocytes are administered every 3-4 weeks, in the absence of GVHD.

After completion of study therapy, patients are followed from engraftment through day 100, and then at 6 months, 1 year, and annually thereafter for 2-5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Langerhans cell histiocytosis (LCH) by demonstration of CD1a positivity or Birbeck granules in lesions
* Considered poor-risk, defined as multisystem disease with involvement of one or more risk organs (i.e., liver, spleen, lungs, and/or hematopoietic system)

  * No isolated "lung only" LCH
* Progressive disease after one of the following treatments:

  * LCH-III protocol or other standard LCH-directed therapies
  * At least 1 course of the current salvage protocol (i.e., LCH-2 2005) or similar therapy (e.g., cytosine arabinoside or cladribine-based regimens)
* HLA-matched related or unrelated donor OR unrelated umbilical cord blood (UCB) available

  * 1 locus mismatch for donor allowed
  * Up to 2 loci mismatch for unrelated UCB allowed
* Any hematologic status (transfusion support allowed)
* Adequate hepatic, renal, cardiac, and pulmonary function to undergo reduced-intensity hematopoietic cell transplantation (RI-HCT) including the following:

  * Transaminases < 5 times upper limit of normal (ULN)
  * Bilirubin < 3 times ULN (unless secondary to hepatic LCH)
  * Creatinine ≤ 2 mg/dL (adults) (if creatinine > 1.2 OR history of renal dysfunction, must have estimated creatinine clearance > 40 mL/min)
  * Creatinine clearance > 40 mL/min (pediatrics)
  * Glomerular filtration rate ≥ 50mL/min
* Negative pregnancy test

Exclusion Criteria:

* Decompensated congestive heart failure, uncontrolled arrhythmia, or left ventricular ejection fraction ≥ 35%
* Pulmonary failure (i.e., requiring mechanical ventilation) unless secondary to active underlying LCH
* Isolated liver sclerosis or pulmonary fibrosis unless secondary to active underlying LCH
* Uncontrolled active life-threatening infection
* Pregnant or nursing
* Less than 4 weeks after last attempted salvage chemotherapy treatment
* Other concurrent chemotherapy agents (e.g., methotrexate) during entire transplantation period up to day 100 post-transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Smith, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Alemtuzumab Conditioning: Patients administered with alemtuzumab, fludarabine phosphate, melphalan and donor stem cell transplantation in children with resistant Langerhans cell histiocytosis.
  alemtuzumab: Administered intravenously (IV) 0.2 mg/kg on Days -8 through -4.
  fludarabine phosphate: Administered 30 mg/m2 intravenously (IV) over 30-60 min on Days -7 through -3.
  (dose adjust if age <12 months)
  melphalan: Administered 140 mg/m2 intravenously (IV) over 30 min on Day -2 (dose adjust if age <12 months)
  stem cell transplantation: Administered as allogeneic hematopoietic, peripheral blood or umbilical cord blood transplantation
Period: Overall Study
Arm/Group | Alemtuzumab Conditioning
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab Conditioning
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Count of patients alive at 1 and 3 years. Deaths from any cause are events. Surviving patients are censored at the date of last contact.
Time Frame: Year 1, Year 3
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Conditioning
Number analyzed (Participants) | 1
participants | 0

2. Primary Outcome: Disease-free Survival at 12 Months Post Transplantation
Description: This outcome is defined as survival with resolution of LCH at 12 months post transplant.
  Unresolved disease for over 12 months post-transplant, progressive disease after this time period, recurrence of disease and death from any cause are considered events.
  Those who survive with resolution of disease are censored at the date of last contact.
Time Frame: Year 1
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Conditioning
Number analyzed (Participants) | 1
participants | 0

3. Secondary Outcome: Transplantation-related Death
Description: Count of patients who died by day 100 related to the transplantation.
Time Frame: Day 100
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Conditioning
Number analyzed (Participants) | 1
participants | 0

4. Secondary Outcome: Neutrophil Engraftment
Description: Incidence of neutrophil recovery and donor chimerism at Day 100.
Time Frame: Day 100
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Conditioning
Number analyzed (Participants) | 1
participants | 1

5. Secondary Outcome: Incidence of Grade II-IV Acute Graft-versus-host-disease (GVHD)
Description: The occurrence of skin, gastrointestinal or liver abnormalities fulfilling the criteria of Grades II, III and/or IV acute GVHD are considered events (Appendix II). Patients without acute GvHD will be censored at the time of death or last follow-up. Patients that survive <21 days and listed as not evaluable will be excluded. Patients receiving a second transplant will be censored at the time of second transplant.
Time Frame: Day 100 and Month 6
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Conditioning
Number analyzed (Participants) | 1
participants | 1

6. Secondary Outcome: Incidence of Chronic GVHD
Description: Occurrence of symptoms in any organ system fulfilling the criteria of limited or extensive chronic GvHD (Appendix III), among patients surviving > 90 days with evidence of engraftment. Patients without chronic GvHD will be censored at time of death or last follow-up.
Time Frame: Day 100 and Month 6
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Conditioning
Number analyzed (Participants) | 1
participants | 0

7. Secondary Outcome: Platelet Engraftment
Description: Incidence of platelet recovery and donor chimerism at Day 100.
Time Frame: Day 100
Measure: Number; unit: participants
Groups:
- Alemtuzumab: Patients administered with alemtuzumab, fludarabine phosphate, melphalan and donor stem cell transplantation in children with resistant Langerhans cell histiocytosis.
  alemtuzumab: Administered intravenously (IV) 0.2 mg/kg on Days -8 through -4.
  fludarabine phosphate: Administered 30 mg/m2 intravenously (IV) over 30-60 min on Days -7 through -3.
  (dose adjust if age <12 months)
  melphalan: Administered 140 mg/m2 intravenously (IV) over 30 min on Day -2 (dose adjust if age <12 months)
  stem cell transplantation: Administered as allogeneic hematopoietic, peripheral blood or umbilical cord blood transplantation
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 1
participants | 0

8. Secondary Outcome: Incidence of Grade III-IV Acute Graft-versus-host-disease (GVHD)
Description: as for outcome 5
Time Frame: Day 100 and Month 6
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Conditioning
Number analyzed (Participants) | 1
participants | 0

ADVERSE EVENTS:
Time Frame: The adverse event data were collected at 100 days post-transplantation.
Arm/Group | Alemtuzumab Conditioning
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab Conditioning (N=1)
Respiratory syncytial virus (RSV) infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab Conditioning (N=1)
Multiple systemic infections (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes